CLINICAL TRIAL: NCT01149876
Title: A Single Blind, Placebo Controlled Trial to Evaluate Effects of a Study Medication, a Nu Skin Lightening Product With and Without Iontophoresis vs Tretinoin Cream vs Vehicle Control for Facial Hyperpigmentation
Brief Title: Study to Evaluate the Effect of a Nu Skin Product and Device for Brown Spots
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Molly A. Wanner, MD, Assistant Physician, Dermatology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-P-002803
Record Dates: First submitted 2010-04-30; First posted 2010-06-24 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nu Skin Product (Experimental)
  Interventions: Other: Nu Skin Product
- Nu Skin product with galvanic spa system (Experimental)
  Interventions: Other: Nu Skin Product; Other: Cosmetic instrument
- Tretinoin cream 0.05 (Active Comparator)
  Interventions: Drug: Tretinoin cream 0.05
- over the counter moisturizer (Placebo Comparator)
  Interventions: Other: CeraVe moisturizer

INTERVENTIONS:
Other: Nu Skin Product — Thin layer of Nu Skin product applied to face.
  Arms: Nu Skin Product; Nu Skin product with galvanic spa system
Other: Cosmetic instrument — Cosmetic instrument with topical Nu Skin product. Thin layer of Nu Skin product applied to face followed by galvanic, used for 3 minutes.
  Arms: Nu Skin product with galvanic spa system
Drug: Tretinoin cream 0.05 — Thin layer of tretinoin applied to face.
  Arms: Tretinoin cream 0.05
Other: CeraVe moisturizer — Thin layer of CeraVe applied to face.
  Arms: over the counter moisturizer

SUMMARY:
The purpose of this study is to determine whether a topical Nu Skin product with or without a galvanic spa device improves brown spots on the face. The Nu Skin product will be compared to an over the counter moisturizer and tretinoin cream.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign informed consent.
* Able to complete study and comply with study procedures.
* Caucasian female ages 25-55.
* Presence of photodamage and lentigines of II-III on the Glogau Photoaging
* Must be willing to avoid laser and light treatments, treatments with filler, chemical peels, microdermabrasion, Botox or any other cosmetic treatment to the face during the duration of the study.
* Must be willing to avoid changing topical moisturizers and cosmetics during the study.
* Able to stop any alpha or beta hydroxy acids, topical retinol or retinoid derivatives, topical antioxidants, or any topical product that may interfere with the study 2 weeks prior to the study.

Exclusion Criteria:

* Cosmetic treatment of face, such as laser or light treatment, filler, Botox, microdermabrasion, or chemical peels 6 months prior to study or during study.
* Current smoker.
* Pregnant, nursing, or planning to become pregnant during study.
* Currently taking drugs including oral retinoids or any other medication with a known clinically significant drug interaction with topical tretinoin.
* Known hypersensitivity to retinoids. History of severe retinoid dermatitis.
* History of substance abuse, mental dysfunction, or other factors limiting ability to cooperate with study.
* Concurrent participation in another clinical study or participation 30 days prior to enrollment that includes exposure to an investigational drug that would interfere with this study.
* Any disease or condition which would interfere with study participation or unduly increase risk.
* Presence of an electrically sensitive support system such as a pacemaker.
* Known history of epilepsy.
* Presence of metal implants or metal braces on teeth.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Wanner, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 2010-2011.
Pre-assignment Details: Wash out period to allow subjects to d/c any topicals that would interfere with study or met exclusion criteria.
Groups:
- Over the Counter Moisturizer: CeraVe Moisturizer
Period: Overall Study
Arm/Group | Nu Skin Product | Over the Counter Moisturizer | Tretinoin Cream 0.05 | Nu Skin Product With Galvanic Spa System
Started | 21 | 20 | 21 | 18
Completed | 20 | 20 | 20 | 18
Not Completed | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proprietary Topical | Placebo | Tretinoin | Proprietary Topical Plus Iontophoresis | Total
Number analyzed (Participants) | 21 | 20 | 21 | 18 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (6.3) | 46.9 (8.3) | 42.3 (8.7) | 49.6 (5.5) | 46.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 21 | 18 | 80
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 21 | 18 | 80
Baseline Hyperpigmentation Score [Mean (Standard Deviation); unit: units on a scale] | 3.7 (1.03) | 3.35 (.93) | 3.3 (1.17) | 3.28 (1.07) | 3.4 (1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hyperpigmentation of the Face
Description: Primary outcome measure will be change in hyperpigmentation of baseline compared to week 16.
  Hyperpigmentation will be measured clinically using a 0-6 scale where 0 is no hyperpigmentation and 6 is very severe hyperpigmentation.
Time Frame: baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Over the Counter Moisturizer: CeraVe cream
Arm/Group | Nu Skin Product | Over the Counter Moisturizer | Tretinoin Cream 0.05 | Nu Skin Product With Galvanic Spa System
Number analyzed (Participants) | 20 | 20 | 20 | 18
units on a scale | .8 (.89) | .3 (.66) | .45 (.69) | .56 (.7)
Statistical Analysis 1: Comparison: Nu Skin Product vs Over the Counter Moisturizer; Test type: Superiority or Other; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Over the Counter Moisturizer vs Tretinoin Cream 0.05; Test type: Superiority or Other; p = .25, t-test, 2 sided
Statistical Analysis 3: Comparison: Over the Counter Moisturizer vs Nu Skin Product With Galvanic Spa System; Test type: Superiority or Other; p = .48, t-test, 2 sided

2. Secondary Outcome: Change in Rhytides
Description: Secondary outcome measures will be change in rhytides of baseline compared to week 16.
  Rhytides will be assessed clinically using a 0-6 scale where 0 is no lines and 6 is very deep lines.
Time Frame: baseline to week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nu Skin Product | Over the Counter Moisturizer | Tretinoin Cream 0.05 | Nu Skin Product With Galvanic Spa System
Number analyzed (Participants) | 20 | 20 | 20 | 18
units on a scale | .25 (.91) | .4 (.75) | -.05 (.69) | .47 (.51)

ADVERSE EVENTS:
Arm/Group | Proprietary Topical | Placebo | Tretinoin | Proprietary Topical Plus Iontophoresis
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 10/21 | 13/20 | 20/21 | 17/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proprietary Topical (N=21) | Placebo (N=20) | Tretinoin (N=21) | Proprietary Topical Plus Iontophoresis (N=18)
Dental Abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GI upset (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low Vit D (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) | 3 (3) | 3 (3)
Tennis elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peeling skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metal taste (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Dryness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HSV (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Mild shock (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pinched nerve (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritant dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VZV (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain with eating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flaking of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angiofibroma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental filling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Scale of pigmentation didn't account for both change in color and number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No